CLINICAL TRIAL: NCT04115059
Title: Dasatinib in Patients With Waldenström Macroglobulinemia (WM) Progressing on Ibrutinib
Brief Title: Dasatinib In Waldenström Macroglobulinemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Jorge J. Castillo, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Jorge J. Castillo, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-305
Record Dates: First submitted 2019-10-02; First posted 2019-10-03 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-09

CONDITIONS: Waldenstrom Macroglobulinemia; DASATINIB
Keywords: Waldenstrom Macroglobulinemia; DASATINIB
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dasatinib (Experimental): -- After the screening procedures confirm participation in the research study: The participant will be given a study drug-dosing calendar for each treatment cycle.
  Dasatinib: Oral Study Drug(s):
  * Each study treatment cycle lasts 4 weeks during which time you will be taking the study drug one time per day.
  * This will continue for up to 24 cycles.
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Oral, daily, dosing per protocol, once a day for cycle
  Other Names: Sprycel

SUMMARY:
This is Phase I pilot, single center study designed to explore the safety of Dasatinib in symptomatic Waldenström Macroglobulinemia participants who are progressing on ibrutinib therapy with BTK Cys481 or PLCG2 mutations

DETAILED DESCRIPTION:
This research study is a Pilot Study, which is the first time investigators are examining this drug in patients with Waldenström Macroglobulinemia who have progressed on ibrutinib.

Patients who fulfill eligibility criteria will be entered into the trial to receive Dasatinib

After the screening procedures confirm participation in the research study:

The participant will be given a study drug-dosing calendar for each treatment cycle. In this research study, the investigators are planning to give Dasatinib, which is a targeted therapy intended to treat cancer by binding to the target protein called BTK.

* BTK is believed to be an important target for treatment of patients with specific gene mutations. Some patients who have disease progression after taking ibrutinib have these gene mutations.
* Making treatment decisions based on genetic testing is investigational, and the FDA has not approved this genetic testing.

The U.S. Food and Drug Administration (FDA) has not approved Dasatinib for Waldenström Macroglobulinemia but it has been approved for other uses.

Dasatinib is produced by Bristol-Myers Squibb.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate. Screening evaluations including consent, physical exam, and laboratory assessments will be done within 30 days prior to Cycle 1 Day 1. Bone marrow biopsy & aspirate, and CT C/A/P will be done within 90 days prior to Cycle 1 Day 1.
* Clinicopathological diagnosis of Waldenstrom's Macroglobulinemia
* Known tumor expression of mutated MYD88 performed by a CLIA certified laboratory.
* Participants must have a BTKCys481 and/or PLCγ2 mutation. Genomic alterations must be confirmed via sequencing performed at NeoGenomics Laboratories
* At least one previous therapy, with ibrutinib as the most recent treatment. Participants may remain on ibrutinib therapy during screening. A 1 day washout before starting dasatinib is required.
* Documented disease progression on last regimen (ibrutinib) per the Sixth International Workshop on WM. One or more of the following:
* 25% increase in serum IgM level with at least 500 mg/dL absolute increase from nadir with re-confirmation
* Progression of clinically significant disease related symptoms
* Symptomatic disease meeting criteria for treatment using consensus panel criteria from the Second International Workshop on WM [26]. One or more of the following:

  * Constitutional symptoms
  * Progressive or symptomatic lymphadenopathy or splenomegaly
  * Hemoglobin <10 g/dL
  * Platelet count <100 k/uL
  * Symptomatic peripheral neuropathy
  * Systemic amyloidosis
  * Renal insufficiency
  * Symptomatic cryoglobulinemia
* Age 18 years or older
* Measurable disease, defined as presence of immunoglobulin M (IgM) paraprotein with a minimum serum IgM level of > 2 times the upper limit normal.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Women of childbearing potential: Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or have or will have complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) while participating in the study; and 2) for at least 28 days after discontinuation from the study. FCBP must be referred to a qualified provider of contraceptive methods if needed.
* Men must agree to use a latex condom during sexual contact with a female of childbearing potential (FCBP) even if they have had a successful vasectomy.
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥500/ uL (Growth factor not permitted)
  * Platelets ≥50,000/ uL (Platelet transfusion not permitted)
  * Hemoglobin ≥ 7 g/dL (RBC transfusion permitted)
  * Total bilirubin ≤ 2 mg/dL
  * Potassium ≥ LLN
  * Magnesium ≥ LLN
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * Estimated GFR ≥ 30 ml/min
* Able to swallow pills.
* Able to adhere to the study visit schedule and other protocol requirements.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study:
* Lactating or pregnant women.
* Participants who are receiving any other investigational agents.
* Prior therapy with BCR-ABL inhibitors.
* Known CNS lymphoma.
* Symptomatic hyperviscosity requiring urgent therapy.
* Human Immunodeficiency Virus (HIV), active infection with Hepatitis B Virus (HBV), and/or Hepatitis C Virus (HCV).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, pleural or pericardial effusion, unstable angina pectoris, cardiac arrhythmia, QT Prolongation, or psychiatric illness/social situations that would limit compliance with study requirements.
* Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec)
* History clinically significant ventricular arrhythmias such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes
* Known history of alcohol or drug abuse
* On any active therapy for other malignancies with the exception of topical therapies for basal cell or squamous cell cancers of the skin.
* History of non-compliance to medical regimens.
* Treatment with strong CYP3A4/5 inhibitors or inducers
* Participants who are taking St. Johns Wort. Must discontinue at least 5 days before starting dasatinib.
* Treatment with H2 Antagonists and proton pump inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Castillo, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Castillo JJ, Sarosiek S, Flynn CA, Leventoff C, Little M, White T, Meid K, Treon SP. A pilot study on dasatinib in patients with Waldenstrom macroglobulinemia progressing on ibrutinib. EJHaem. 2022 Jun 7;3(3):927-929. doi: 10.1002/jha2.493. eCollection 2022 Aug. PMID 36051045

RESULTS

PARTICIPANT FLOW:
Groups:
- Dasatinib: -- After the screening procedures confirm participation in the research study: The participant will be given a study drug-dosing calendar for each treatment cycle.
  Dasatinib: Oral Study Drug(s):
  * Each study treatment cycle lasts 4 weeks during which time you will be taking the study drug one time per day.
  * This will continue for up to 24 cycles.
  Dasatinib: Oral, daily, dosing per protocol, once a day for cycle
Period: Overall Study
Arm/Group | Dasatinib
Started | 3
Completed | 0
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 73 [46 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Treatment-Emergent Adverse Event
Description: Count of participants who experience a treatment-emergent adverse event
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 3
Participants | 3

2. Secondary Outcome: Overall Response Rate
Description: Percentage of patients with an Overall Response. Overall Response Rate= Minor response (>25%-50% reduction in serum IgM from baseline) + Partial Response (>50-90% reduction in serum IgM from baseline) + Very Good Partial Response (>90% reduction in serum IgM from baseline) + Complete Response (resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 3
Participants | 0

3. Secondary Outcome: Complete Response Rate
Description: Percentage of patients with Complete Response (CR). Complete Response requires resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, and resolution of any adenopathy or splenomegaly.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 3
Participants | 0

4. Secondary Outcome: Very Good Partial Response Rate
Description: Percentage of patients with very good partial response (VGPR) to therapy. (VGPR is >90% reduction in serum IgM from baseline)
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 3
Participants | 0

5. Secondary Outcome: Partial Response Rate
Description: Percentage of patients with partial response (PR) to therapy. (PR is 50-89% reduction in serum IgM from baseline)
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 3
Participants | 0

6. Secondary Outcome: Minimal Response Rate
Description: Percentage of patients with Minor Responses to therapy. (MR is 25-49% reduction in serum IgM from baseline)
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 3
Participants | 0

7. Secondary Outcome: Stable Disease Rate
Description: Percentage of patients with Stable disease to therapy. (SD is <25% reduction in serum IgM from baseline).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 3
Participants | 3

8. Secondary Outcome: Progressive Disease Rate
Description: Percentage of patients with who experienced disease progression on study. PD is >25% increase in serum IgM from baseline with an absolute increase of at least 500 mg/dL, or progression of clinically significant disease related symptoms. Death from any cause or initiation of a new anti-neoplastic therapy will also be considered a progression event. An increase of 1 cm in any axis for adenopathy, or 2 cm in the craniocaudal axis of the spleen will be considered evidence of progression of extramedullary disease. Development of Bing Neel syndrome, or other extramedullary disease manifestations, as well as disease transformation will be considered as progressive events.
Time Frame: From first dose through disease progression, up to 2 years from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 3
Participants | 2

9. Secondary Outcome: Progression Free Survival
Description: The amount of time between starting treatment and experiencing disease progression. PD is >25% increase in serum IgM from baseline with an absolute increase of at least 500 mg/dL, or progression of clinically significant disease related symptoms. Death from any cause or initiation of a new anti-neoplastic therapy will also be considered a progression event. An increase of 1 cm in any axis for adenopathy, or 2 cm in the craniocaudal axis of the spleen will be considered evidence of progression of extramedullary disease. Development of Bing Neel syndrome, or other extramedullary disease manifestations, as well as disease transformation will be considered as progressive events.
Time Frame: From first dose through disease progression, up to 2 years from baseline
Measure: Median (Full Range); unit: months
Arm/Group | Dasatinib
Number analyzed (Participants) | 3
months | 5 [0 to 5]

10. Secondary Outcome: Time to Next Therapy (TTNT)
Description: The amount of time between starting study treatment and initiating a new therapy
Time Frame: From first dose through initiation of new therapy, up to 2 years from baseline
Measure: Median (Full Range); unit: months
Arm/Group | Dasatinib
Number analyzed (Participants) | 3
months | 6 [1 to 6]

11. Secondary Outcome: Overall Survival
Description: The number of participants who are still alive at the end of follow-up. Participants were observed for up to 2 years after discontinuing study therapy for survival status.
Time Frame: From first dose through death, up to 2 years from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 3
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected after dasatinib initiation, through 30 days after the last dose of dasatinib (e.g. 6 months). Participants were observed for overall survival for up to 2 years, or until withdrawal of consent or death.
Arm/Group | Dasatinib
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=3)
Metapneumovirus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (3)
Arrhythmia (Cardiac disorders) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=3)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Congestive heart failure (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Abdominal distention (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Mouth sores (Gastrointestinal disorders) | 1 (1)
Edema (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Fluid overload (General disorders) | 1 (1)
Leg edema (General disorders) | 1 (1)
Withdrawal symptoms (General disorders) | 1 (1)
Neutropenia (Investigations) | 1 (1)
Thrombocytopenia (Investigations) | 1 (1)
Body Aches (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Migraines (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT04115059/Prot_SAP_000.pdf